CLINICAL TRIAL: NCT07214025
Title: Safety and Efficacy of Romiplostim in Treatment of Chronic ITP in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Refat Mostafa Ali, Principal Investigator, Assiut University
Other Study IDs: Romiplostim In treatmentof ITP
Record Dates: First submitted 2025-09-26; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Romiplostim N01; ITP
MeSH Terms: interventions — Safety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Safety and efficacy of Romiplostim in Treatment of chronic ITP in children — Children diagnosed with chronic immune thrombocytopenia (ITP) will receive Romiplostim, a thrombopoietin receptor agonist administered as a once-weekly subcutaneous injection. The initial dose will be 1 µg/kg, with subsequent dose adjustments (up to a maximum of 10 µg/kg weekly) based on platelet response, in order to maintain platelet counts ≥50 × 10⁹/L while minimizing the risk of bleeding. Treatment duration will be determined according to study protocol, and patients will be monitored regularly for efficacy (platelet count response, bleeding events) and safety (adverse events, laboratory parameters).

SUMMARY:
The aim is to evaluate safety and efficacy of Romiplostim in the treatment of chronic ITP in children

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 1 and 18 years
* Diagnosis of chronic ITP
* Refractory to or intolerant of first-line therapies (e.g.corticosteroids , intravenous immunoglobulin [ IVIG ] , and oral eltrombopag )
* Platelet count<30,000/µL, or evidence of bleeding or risk of bleeding with platelet count<50,000/µL.
* Written informed consent (or parental/guardian consent for minors)

Exclusion Criteria:

* Evidence of secondary thrombocytopenia (e.g., HIV, HCV, systemic lupus erythematosus)
* congenital thrombocytopenia
* Age < 1year or more than 18 years
* Aplastic anemia
* Known hypersensitivity to romiplostim or any of its components

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include pediatric patients aged 1 to 18 years with a diagnosis of chronic immune thrombocytopenia (ITP) who are refractory to or intolerant of first-line therapies (e.g., corticosteroids, intravenous immunoglobulin, or oral eltrombopag). Eligible patients must have a platelet count <30,000/µL, or evidence of bleeding/risk of bleeding with platelet count <50,000/µL. Patients with secondary or congenital thrombocytopenia, aplastic anemia, age <1 year or >18 years, or known hypersensitivity to romiplostim will be excluded. A total of 100 patients will be enrolled from the Pediatric Department at Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Durable Platelet Response in Patients Receiving Treatment for Chronic ITP | Up to 48 weeks of treatment
  The proportion of patients achieving a durable platelet response, defined as platelet counts ≥50 × 10⁹/L for at least 6 of the final 8 weeks of a 48-week treatment period, without the need for rescue therapy (e.g., IVIG, corticosteroids, platelet transfusion).

SECONDARY OUTCOMES:
Time to Initial Platelet Response | Up to 48 weeks of treatment.
  Time (in days) from initiation of Romiplostim therapy to the first platelet count ≥50×10⁹/L without rescue medication in the preceding 7 days.
Need for Rescue Medications | Up to 48 weeks of treatment.
  Proportion of patients requiring administration of rescue medications (e.g., corticosteroids, intravenous immunoglobulin) during Romiplostim therapy.
Rate of Treatment-Free Remission | Up to 48 weeks of treatment.
  Proportion of patients who maintain platelet counts ≥50×10⁹/L for at least 24 consecutive weeks after discontinuation of Romiplostim without rescue therapy.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Result] Chen F, McDonald V, Newland A. Experts' review: the emerging roles of romiplostim in immune thrombocytopenia (ITP). Expert Opin Biol Ther. 2021 Nov;21(11):1383-1393. doi: 10.1080/14712598.2021.1960979. Epub 2021 Aug 12. PMID 34313512
- [Result] Vianelli N, Auteri G, Buccisano F, Carrai V, Baldacci E, Clissa C, Bartoletti D, Giuffrida G, Magro D, Rivolti E, Esposito D, Podda GM, Palandri F. Refractory primary immune thrombocytopenia (ITP): current clinical challenges and therapeutic perspectives. Ann Hematol. 2022 May;101(5):963-978. doi: 10.1007/s00277-022-04786-y. Epub 2022 Feb 24. PMID 35201417
- [Result] Liu XG, Hou Y, Hou M. How we treat primary immune thrombocytopenia in adults. J Hematol Oncol. 2023 Jan 19;16(1):4. doi: 10.1186/s13045-023-01401-z. PMID 36658588
- [Result] Singh A, Uzun G, Bakchoul T. Primary Immune Thrombocytopenia: Novel Insights into Pathophysiology and Disease Management. J Clin Med. 2021 Feb 16;10(4):789. doi: 10.3390/jcm10040789. PMID 33669423
- [Result] Sandvad M, Pedersen EA, Frederiksen H, Mannering N. Risk of infection in adult patients with primary immune thrombocytopenia (ITP): a systematic review. Expert Rev Hematol. 2021 Oct;14(10):961-974. doi: 10.1080/17474086.2021.1976635. Epub 2021 Sep 16. PMID 34487679